CLINICAL TRIAL: NCT01117935
Title: Study of Hypofractionated Intensity Modulated External Beam Therapy for the Treatment of Patients With Adenocarcinoma of the Prostate
Brief Title: Intensity-Modulated External Beam Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-12870; NCI-2010-00877 (Registry Identifier: CTRP)
Record Dates: First submitted 2010-04-30; First posted 2010-05-06 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Adenocarcinoma of the Prostate; Stage I Prostate Cancer; Stage II Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
Keywords: IMRT; prostate cancer; radiation therapy; external beam; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm I (Experimental): Patients undergo hypofractionated intensity modulated radiotherapy once daily, 5 days a week, for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients with intermediate- and high-risk disease may also receive concurrent and adjuvant or long-term androgen deprivation therapy for up to 36 months.
  Interventions: Radiation: intensity modulated external beam radiation therapy

INTERVENTIONS:
Radiation: intensity modulated external beam radiation therapy — Low risk - 69.6 Gy in 2.4 Gy fractions to prostate
  Intermediate risk - delivered in 30 fractions with neoadjuvant and concurrent androgen deprivation therapy: 72 Gy in 2.4 Gy fractions to prostate + 60 Gy in 2 Gy fractions to seminal vesicles +/- 50.4 Gy in 1.68 Gy fractions to lymph nodes
  High risk - 30 fractions with neoadjuvant, concurrent, and long term adjuvant androgen deprivation therapy: 72 Gy in 2.4 Gy fractions to prostate + 60 Gy in 2 Gy fractions to seminal vesicles +/- 50.4 Gy at 1.68 Gy fractions to lymph nodes
  Other Names: EBRT; IMRT

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. Specialized radiation therapy, such as intensity-modulated radiation therapy, that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This clinical trial studies intensity-modulated external beam radiation therapy in treating patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate that patients can safely receive IMRT teletherapy using the proposed IMRT fractionation schedule without experiencing a treatment limiting toxicity.

SECONDARY OBJECTIVES:

I. To assess treatment efficacy through the surrogate measures of PSA nadir and biochemical failure-free survival.

OUTLINE: Patients undergo hypofractionated intensity modulated radiotherapy once daily, 5 days a week, for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients with intermediate- and high-risk disease may also receive concurrent and adjuvant or long-term androgen deprivation therapy for up to 36 months. After completion of study treatment, patients are followed at 4-6 weeks, every 4 months for 3 years, every 6 months for 2 years, and then annually until year 5.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven adenocarcinoma of the prostate are eligible for protocol enrollment when the following criteria are met; patients must have low, intermediate or high-risk adenocarcinoma of the prostate, as defined by the National Comprehensive Cancer Network (NCCN) criteria
* A diagnostic CT scan of the abdomen and pelvis will be obtained to rule out regional disease (maximum of 60 days prior to registration) for high-risk patients only
* A bone scan showing no evidence of metastatic disease is also required for patients whose prostate-specific antigen (PSA) is greater than 20 ng/ml, Gleason's sum is greater than 7, or T-stage is greater than T2b
* Alkaline phosphatase within 1.5 x upper limit of normal (ULN) is required for all patients beginning hormone therapy
* AST within 1.5 x ULN is required for all patients beginning hormone therapy
* Bilirubin within 1.5 x ULN is required for all patients beginning hormone therapy
* Karnofsky Performance score >= 80
* Prior to registration, patients having received no more than three months treatment with anti-androgen, luteinizing hormone-releasing hormone (LHRH) agonist, or a combination of the two remain eligible for protocol treatment; the qualifying PSA for these patients will be the value recorded prior to the initiation of the hormone therapy

Exclusion Criteria:

* Patients with history of inflammatory bowel disease, or who require steroid or cytotoxic therapy for collagen vascular disease
* Patients with a history of cancer other than skin cancer within five years of the initiation of protocol treatment
* Patients with a history of pelvic irradiation for any reason

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-05-30; Primary Completion 2015-06-25 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Toxicity as measured by Common Terminology Criteria for Adverse Events (CTCAE) v3 criteria | At 2 years

SECONDARY OUTCOMES:
Biochemical failure as defined by the Phoenix definition | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael G. Chang, MD, Principal Investigator — Massey Cancer Center
Locations (2):
- United States (2):
  - Hunter Holmes McGuire Veterans Administration Medical Center, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Derived] Ricco A, Mukhopadhyay N, Deng X, Holdford D, Skinner V, Saraiya S, Moghanaki D, Anscher MS, Chang MG. Moderately Hypofractionated Intensity Modulated Radiation Therapy With Simultaneous Integrated Boost for Prostate Cancer: Five-Year Toxicity Results From a Prospective Phase I/II Trial. Front Oncol. 2020 Aug 21;10:1686. doi: 10.3389/fonc.2020.01686. eCollection 2020. PMID 32974208
- See also: VCU Massey Cancer Center — http://www.massey.vcu.edu/